CLINICAL TRIAL: NCT06882629
Title: The Effect of Virtual Reality Homework Exercises As an Add-On to Behavioral Therapy for Children with Selective Mutism
Brief Title: VR Homework Exercises for Selective Mutism Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luuk Stapersma (Other)
Responsible Party: Sponsor-Investigator, Luuk Stapersma, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL86645.018.24
Record Dates: First submitted 2025-02-04; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Selective Mutism; Anxiety Disorder of Childhood
Keywords: Virtual reality; Virtual reality exposure therapy; Intervention; Treatment; Children; Anxiety
MeSH Terms: conditions — Mutism; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Behavioral: 'Speaking at school, a matter of doing' combined with VR homework exercises
  Interventions: Behavioral: 'Speaking at school, a matter of doing' combined with VR homework exercises

INTERVENTIONS:
Behavioral: 'Speaking at school, a matter of doing' combined with VR homework exercises — The treatment in this study consists of behavioral therapy for selective mutism (with the protocol 'Speaking at school, a matter of doing') with the addition of the VR homework exercises. The protocol consists of 10 steps that help the child to gain confidence while speaking at school. For every treatment step there are VR homework exercises available. Families receive a VR headset for the duration of the study. Parents are instructed to work on the VR homework exercises at least once a week and encouraged to work on the VR homework exercises several times a week.

SUMMARY:
Selective mustism (SM) is an anxiety disorder that manifests in childhood. Children with Children with SM do not speak in certain social situations where this is expected of them. For example, a child may talk at home, but is afraid to speak at school. The goal of this clinical trial is to determine the efficacy of behavioral therapy for children with selective mutism (SM) combined with virtual reality (VR) homework exercises. Virtual Reality Exposure is an effective treatment for adults with anxiety disorders.

The main questions to answer are:

* Is behavioral therapy combined with VR homework exercises effective in the treatment of SM?
* Which familial factors contribute to a positive treatment outcome and homework adherence?

A single-case experimental design (SCED) will be used to evaluate the efficacy of the treatment. The child's speaking behavior at baseline will be compared to the child's speaking behavior in the different phases of the intervention.

Participants will:

* Follow individual therapy sessions at school.
* Practice with the VR homework exercises at least once a week.
* Parents and teachers will evaluate the child's speaking behavior.

DETAILED DESCRIPTION:
The treatment in this study consists of behavioral therapy for SM (with the protocol 'Talking at school, a matter of doing') with the addition of the VR homework exercises. The protocol consists of 10 steps that help the child to gain confidence while speaking at school. The individual therapy sessions are provided at school. For every step of the protocol there are VR homework exercises available. Families receive a VR headset for the duration of the study. Parents are instructed to work on the VR homework exercises at least once a week and encouraged to work on the VR homework exercises several times a week. On average, treatment is approximately 25 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The child meets the DSM-5 criteria for SM (as a primary classification).
* The child is attending primary school.
* Referred to an academic center for Child and Adolescent Psychiatry (Levvel) for diagnosis and treatment of SM
* Psychiatric comorbidity is permitted, given that SM is the primary treatment target.
* Medication use is permitted, if stable for at least 4 weeks prior to the start of treatment.

Exclusion Criteria:

* No participating parents.
* Parents do not have sufficient mastery of the Dutch language.
* Parents or child have an estimated IQ below 75.
* The child needs inpatient treatment.
* Children with a (medical) condition that is a contraindication for using a VR headset (epilepsy, claustrophobia, facial condition, sensitive vestibular system, panic attacks)
* Parents receiving parental guidance which is not part of the standard treatment program.
* Children that have received protocolled behavior therapy for SM in the past 12 months.

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
SM symptoms (frequent measurement) | During the baseline period (2 weeks), during the intervention phase (up to 1 year) and during follow-up (3 months after end of intervention phase), three times a week
  Both parents and teachers are asked to report on SM symptoms. This is done by answering 9 yes/no questions on the child's speaking behavior and communication, including non-verbal communication, making sounds and conversing with others (more yes indicates more speaking behavior). The short assessment is specifically designed for this study in collaboration with experienced SM therapists and a statistician, specialized in SCED's.
SM symptoms (SMQ-NL) | Baseline (2 weeks), start first phase of intervention (up to 4 months), start second phase of intervention (up to 4 months), start training phase, immediately after intervention (up to 4 months), at follow-up (3 months after end of intervention)
  Evaluated by parents. The SMQ consists of 23 questions that are scored on a 4-point Likert scale ranging from "always" to "never." The symptom subscale consists of 17 questions (0-68; higher scores indicate more SM symptoms), that assess the severity of the symptoms across different situations (family, school and public situations). The second subscale indicates to what extend a child experiences problems due to not speaking in certain situations.
SM symptoms (Social context of speaking) | Baseline (2 weeks), start first phase of intervention (up to 4 months), start second phase of intervention (up to 4 months), start training phase (up to 4 months), immediately after intervention, at follow-up (3 months after end of intervention)
  The questionnaire consists of 16 questions assessing (0-64; higher scores indicate less SM symptoms) the social context of speaking assesses the severity of symptoms at school across different social situations (e.g. their own teacher, another teacher, in the classroom or in the presence of peers), speaking behaviour (e.g. whispering and functional speech) and its interference at school. Teachers are asked to evaluate how often child is showing different speaking behaviours and in which social context on a 4-point Likert scale. The questionnaire includes 8 questions that are based on the School Speech Questionnaire (SSQ). For the purpose of our study, the SSQ does not provide enough detail on the child's speaking behaviour, for that reason 8 more questions were included.

SECONDARY OUTCOMES:
VR data | During intervention phase (up to 1 year; every time child uses the VR homework exercises at home)
  Each parent has a unique ID to sign-in to a web-based application that is used to guide the child through the virtual school. Parents will indicate that when the next exercise is presented. These responses are saved. Every time the parent signs in, the total time and the time spent playing the different games will be automatically stored on a secured database. This will be recorded in seconds.
VR completion | During the intervention phase (once a week, up to 1 year)
  Parents are asked to track the time they spend working on the VR homework exercises on a VR tracking sheet on a weekly basis. They are asked to fill out how long and which days they practiced. The number of days practiced will be divided by the total number of days in the week. This yields a percentage of VR completion per week.
VR immersion | During the intervention phase (once a month, up to 1 year)
  Specifically for this study three questions were designed to measure the level of immersion children experience while practicing with the VR. Children are asked to rate their immersive experience on 4-point Likert scale ranging from strongly disagree to strongly agree.
Structured Clinical Interview for DSM-5 Junior (SCID-5-Junior) | Baseline (2 weeks), immediately after intervention (up to 1 year) and at follow-up (3 months after end of intervention)
  Semi-structured interview for children and adolescents between 8 -18. The interview is suitable for both children and their parents. The SCID-5 Junior consists of 17 modules to classify DSM-5 disorders. The SCID-5 Junior is used in standard clinical care, to check for additional anxiety disorders and disorders that might look like SM. The SCID-5 Junior will be administered in the same manner as in regular clinical care, meaning that parents only report on the modules: anxiety, autism and obsessive-compulsive behavior, unless there are indications that suggest the presence of another co-morbid disorder.
Fear Survey Schedule for Children - Revised (FSSC-R or in Dutch VAK 4-12) | Baseline (2 weeks), immediately after intervention (up to 1 year) and at follow-up (3 months after end of intervention)
  The FSSC-R / VAK 4-12 is a self-report questionnaire that consists of 80 items (0-240; higher scores indicate more anxiety symptoms). The items are descriptions of objects or situations that may cause anxiety. The questionnaire can be administered verbally for children who are not able to read. Children are asked to indicate for each item whether it makes them feel 'not anxious', 'a little bit anxious' or 'very anxious'.
Child Behaviour Checklist (CBCL) | Baseline (2 weeks), immediately after intervention (up to 1 year) and at follow-up (3 months after end of intervention)
  The CBCL aims to quantify problem behavior and competences of children and adolescents. This questionnaire with 113 items (0-226, higher scores indicate more emotional and behavioral problems) is used in standard clinical care for routine outcome measuring. The questionnaire is filled out by the parents or caregivers of the child. Parents (both mothers and fathers) indicate on a 3-point scale whether the behavior was present in the last few months. The behavior can be classified according to different scales: Internalizing, Externalizing and other problems.
Teacher Report Form (TRF) | Baseline (2 weeks), immediately after intervention (up to 1 year) and at follow-up (3 months after end of intervention)
  (C-)TRF is the teacher's version of the CBCL. The TRF has 113 items (0-226, higher scores indicate more emotional and behavioral problems) and is included in standard clinical care for routine outcome measuring. The questionnaire can be filled out by a teacher. The questionnaire gives insight in the child's behavior and competences at school as evaluated by the teacher.
Parenting burden questionnaire (OBVL) | Baseline (2 weeks), immediately after intervention (up to 1 year) and at follow-up (3 months after end of intervention)
  With the Dutch OBVL, parents are asked to evaluate statements on how they experience their child and rearing, how they relate to their child and how they are feeling. On a 4-point scale parents indicate to what extend they agree with each statement (34 items, 34-136, higher scores indicate less parenting burden). The OBVL consists of 5 subscales: problems in the caregiver-child relationship, problems with upbringing, depressive moods, role restriction and health problems.
Family Accommodation Scale - Anxiety (FASA) | Baseline (2 weeks), immediately after intervention (up to 1 year) and at follow-up (3 months after end of intervention)
  The questionnaire evaluates the level of family accommodation related to the child's anxiety and the level of distress the child experiences. The FASA consists of 13-questions that are scored on a 5-point Likert scale ranging from "never" to "daily". The first 9 items form the total accommodation scale (0-36, higher scores indicate more family accommodation). The subscale assessing the level of distress (5 items) is scored on a 5-point Likert scale ranging from "no" to "extreme." The FASA is included in standard clinical care for routine outcome measuring.
Clinical global impression of outcome (CGI) | During the intervention phase (up to 1 year), at the end of every therapy session with therapist
  The CGI is a 2-item, clinician-rated scale used to assess global illness severity (1-7; higher score indicates more severity), over-all improvement (1-7, higher score indicates less improvement) from the start of treatment.
Outcome Rating Scale (ORS) | During the intervention phase (up to 1 year), at the end of every therapy session with therapist
  The Outcome Rating Scale (ORS) is used to monitor children's, young people and their families' or caregivers' feedback on therapeutic progress. The ORS is a 4-item session-by-session measure designed to assess areas of life functioning known to change as a result of therapeutic intervention. These areas include: personal or symptom distress, interpersonal well-being, social role and overall well-being (for each item 0-10; higher scores indicate better functioning)
Therapy evaluation: Visual Facial Anxiety Scale (VFAS) | During the intervention (up to 1 year; at the end of each VR session at home and at the end of each therapy session with therapist)
  Children are asked to indicate the level of anxiety, using a visual analogue scale, after completing a VR session and after individual therapy. The child can indicate whether they feel none, mild, mild - moderate, moderate, moderate - high or high anxiety.
Qualitative interview child | Immediately after intervention (up to 1 year)
  A qualitative evaluation will be made after the intervention. During the interview the child will be asked to answer a few short semi-structured questions on their experiences with the VR homework exercises.
Monthly VR evaluation | During the intervention (once a month, up to 1 year)
  The researcher will schedule a 15-minute semi-structured interview to ask parents about their experiences during the VR sessions. The interview contains questions re-garding the practical use of the VR headset, how often parents have practised, the level of anxiety their child experiences while practicing and whether their child likes working with the VR homework exercises. Lastly, parents are asked whether there have been any special events that might have had an influence on the child's SM symptoms or the VR sessions.
Qualitative interview parents | Immediately after intervention (up to 1 year), and at follow-up (3 months after the end of the intervention)
  A qualitative evaluation will be made after the intervention and after 3 months of follow-up. Both parents or caregivers are asked to share their experiences with the VR homework exercises and their vision on how the use of the VR homework exercises has helped their child to gain the confidence to speak at school.
Qualitative interview therapists | Immediately after intervention (up to 1 year)
  After the intervention, therapists are asked to share their perspective about the use of the VR homework exercises in addition to the standard treatment. They are asked to identify what factors, such as the relationship with parents or specific characteristics of the child/family contribute or hinder successful usage of the VR homework exercises.

OTHER OUTCOMES:
Adult Self Report (ASR) | Baseline (2 weeks)
  The ASR is a self-report questionnaire for adults (ages 18-59) assessing aspects of adaptive functioning and problems. The questionnaire provides a Total score (123 items, 0-252, higher scores indicate more behavioral and emotional problems) and scores for an Internalizing and Externalizing subscale.
EMBU-P | Baseline (2 weeks)
  The EMBU-P (with the Swedish name Egna Minnen Beträffende Uppfostran - Parent version) rates the parents' own rearing behavior with their children. Rearing behavior is scored on across 4 dimensions: Rejection, Emotional Warmth, Control Attempts and Favoring Subject. It has 83 items (higher scores per dimension indicate more of that rearing behavior, which can be positive or negative).
Communication - Vineland-3-NL | Baseline (2 weeks)
  This questionnaire evaluates adaptive behavior on five domains: communication, daily living skills, socialization, motor skills and maladaptive behavior. The questionnaire is suitable for both parents and teachers. Only the domain communication will be assessed as the presence of speech and language problems is often linked to SM.
Immersive Tendencies Questionnaire - Parent report | Baseline (2 weeks)
  For the purpose of this study, the questions were rephrased to turn the original questionnaire into a parent-report. Parents are asked to evaluate their child's immersive tendencies on a 7-point likert scale, ranging from strongly disagree to strongly agree (10 items, 0-70, higher scores indicate more immersive tendencies).
Intake questionnaire | Baseline (2 weeks), immediately after intervention (up to 1 year) and at follow-up (3 months after the end of the intervention)
  This questionnaire contains questions with regards to background information about the child and his or her family. Questions concerning sex, age, ethnicity, family composition, parental work situation and education level and medical history (including treatment background and earlier diagnoses given to both parents and child) are included.

CONTACTS AND LOCATIONS:
Locations (1):
- Levvel, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No